CLINICAL TRIAL: NCT02522052
Title: Mussels, Inflammation and Rheumatoid Arthritis (MIRA)
Acronym: MIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MIRA
Record Dates: First submitted 2015-04-29; First posted 2015-08-13 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blue mussel diet (Experimental): 5 meals a week including blue mussels
  Interventions: Other: Blue mussel diet
- Meat/control diet (Active Comparator): 5 meals a week including meat
  Interventions: Other: Meat/Control diet

INTERVENTIONS:
Other: Blue mussel diet — 5 meals a week containing blue mussels
  Arms: Blue mussel diet
Other: Meat/Control diet — 5 meals a week containing meat
  Arms: Meat/control diet

SUMMARY:
Rheumatoid arthritis (RA) is a chronic disease that affects ~1% of the population. A large proportion of patients with established disease have persistent high disease activity in spite of existing effective pharmacological treatment. Improved treatment is thus urgently needed, including alternative treatments in addition to optimal pharmacological therapy. The main purpose of this study is to investigate if a high intake of blue mussel (Mytilus Edulis) could decrease inflammation and disease activity in patients with established RA. A secondary goal is to identify novel biomarkers for blue mussel intake and metabolic responses to this diet, using a metabolomics approach with high sensitivity and specificity. A third goal is to look at genetic polymorphisms in relation to long chain polyunsaturated fatty acids (LCPUFA) and inflammatory markers.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic disease that affects ~1% of the population. A large proportion of patients with established disease have persistent high disease activity in spite of existing effective pharmacological treatment. Improved treatment is thus urgently needed, including alternative treatments in addition to optimal pharmacological therapy. The main purpose of this study is to investigate if a high intake of blue mussel (Mytilus Edulis) could decrease inflammation and disease activity in patients with established RA. A secondary goal is to identify novel biomarkers for blue mussel intake and metabolic responses to this diet, using a metabolomics approach with high sensitivity and specificity. A third goal is to look at genetic polymorphisms in relation to LCPUFA and inflammatory markers.

Diet and lifestyle are associated with chronic diseases such as cardiovascular diseases, cancer and diabetes. Here, evidence based dietary treatment guidelines are available. In contrast, for inflammatory diseases such as RA no dietary guidelines exist, reflecting the ambiguous evidence base. Many dietary components are related to the human immune system or to inflammation. Some are co-factors in immune- or inflammatory response, such as zinc. Others are antioxidants, eg selenium, vitamins E and C. RA has been associated with low serum concentrations of zinc, selenium, vitamins D and B6 although some of this may reflect inflammatory response. Dietary effects on RA symptoms have been reported for long chain fatty acids from fish and probiotics have shown to improve function in RA patients. As prebiotics reduce inflammation in other conditions, it may have positive effects also on RA. Most research on antioxidants has focused on single nutrients but a few dietary trials also have been conducted with mixed results. In sum, high-quality studies evaluating the effect of a combination of food items with indicative effects on RA are needed.

Blue mussels are rich in vitamins (B2 and B12) and minerals (iron, selenium and zinc) and contain the LCPUFA eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA).

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-40 kg/m2,
* disease duration >2 years,
* DAS28 >3.0

Exclusion Criteria:

* other Life-threatening disease,
* pregnant,
* lactating,
* food intolerant or allergic to food included in the study.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
difference between disease activity score 28 (DAS28) after the diets | after 11 week intervention
  Measured clinically

SECONDARY OUTCOMES:
difference in inflammatory markers/cytokines (IL-1beta, IL-6, Tumor Necrosis Factor-alfa, IL-10) after the diets | after 11 week intervention
  measured in blood
Difference in Quality of life and health by SF36, EQ5D och HAQ after the diets | after 11 week intervention
  Measured by validated instruments (SF36, EQ5D och HAQ)
Differences and changes in metabolites after the two diets | after 11 week intervention
  Metabolomics Nuclear magnetic resonance (NMR) analysis of serum and urin samples.

OTHER OUTCOMES:
Difference in plasma and RBC fatty acids after the diets and changes during the diets | after 11 week intervention
  Fatty acids in plasma and red blood cells (RBC)
Differences between blood lipids (TAG, HDL, LDL) after the diets | after 11 week intervention
  Serum analysis of TAG, HDL, LDL
Differences in Hb after the diets | after 11 week intervention
  Blood status (Hb)
Eular response criteria | after 11 week intervention
  To interpret effects on DAS28
Stable isotopes in hair | after 11 week intervention
  stable isotopes

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Lindqvist, PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Not in US/Canada, Sweden

IPD SHARING:
Plan to Share IPD: No
Not approved by the Ethical Review board